CLINICAL TRIAL: NCT01154244
Title: Insulin Resistance as Primary Pathogenesis in Newly Diagnosed, Drug naïve Type 2 Diabetes Patients in Korea
Acronym: SURPRISE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Other Study IDs: 113417
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin resistance; Insulin deficiency; HOMA-IR; Drug naive; Diabetes mellitus, type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug naive type II DM: Newly diagnosed type II Diabetes Mellitus
  Interventions: Other: HOMA-IR

INTERVENTIONS:
Other: HOMA-IR — Blood sampling for HOMA-IR and HbA1C, fasting glucose, C-peptide, Lipid profile

SUMMARY:
The purpose of this study is investigating the clinical characteristics of newly diagnosed, drug naïve type 2 diabetic patients according to insulin secretion and insulin resistance.

DETAILED DESCRIPTION:
Primary Objective:To investigate whether insulin resistance or insulin deficiency is primary in the pathogenesis of type 2 diabetes mellitus in Korea Secondary Objectives:To investigate proportion of patients with severe insulin deficiency at diagnosis,To investigate proportion of metabolic syndrome in patients with newly diagnosed, drug-naïve type 2 diabetes mellitus,To investigate proportion of obesity in patients with newly diagnosed, drug-naïve type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:Newly diagnosed, drug naïve type 2 DM patients who gave informed consent, Diagnosis of type 2 DM will be made according to ADA guideline 2009 Exclusion Criteria:Patients age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed Type II DM, Drug naive
Sampling Method: Probability Sample
Enrollment: 1439 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
insulin resistance assessed using HOMA-IR | within 3months after DM diagnosis

SECONDARY OUTCOMES:
proportion of patients with severe insulin deficiency assessed using C-peptide | within 3months after DM diagnosis
proportion of metabolic syndrome in patients | within 3months after DM diagnosis
proportion of obesity in patients | within 3months after DM diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- South Korea (2):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Seoul